CLINICAL TRIAL: NCT07043556
Title: Assessment of Artificial Intelligence Algorithms for ROTEM Analysis in Coagulation Management
Brief Title: Assessment of Artificial Intelligence Algorithms for ROTEM
Status: Recruiting | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, BURHAN DOST, Associated Proffessor, Ondokuz Mayıs University
Other Study IDs: ROTEM-AI
Record Dates: First submitted 2025-06-21; First posted 2025-06-29 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Coagulopathy
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Artificial Intelligence-Based ROTEM Interpretation — A structured artificial intelligence-based evaluation system that analyzes ROTEM (Rotational Thromboelastometry) parameters and provides treatment recommendations. ROTEM case data are converted into standardized clinical scenarios and evaluated by AI models using a predefined template. The AI output is compared to the consensus of expert clinicians regarding the presence and type of coagulopathy and the need for therapeutic intervention (e.g., fibrinogen, protamine, platelets, PCC, plasma). This intervention does not involve any patient-facing activity and is performed on de-identified data only.

SUMMARY:
The goal of this observational validation study is to evaluate whether artificial intelligence (AI) models can accurately interpret ROTEM (Rotational Thromboelastometry) data and provide appropriate treatment recommendations in adult patients undergoing elective cardiac or liver transplantation surgery.

The main questions it aims to answer are:

Can AI models (e.g., ChatGPT and Gemini ) accurately determine whether treatment is indicated based on ROTEM parameters? Can AI models correctly identify the type of coagulopathy (e.g., fibrinogen deficiency, platelet dysfunction)? Are the treatment recommendations from AI models concordant with expert clinical consensus? Researchers will compare the decisions made by AI models to a gold standard expert panel to see if AI models can match or approximate expert-level decision-making in interpreting ROTEM outputs.

Participants will:

Undergo elective cardiac or liver transplant surgery. Have standard ROTEM tests performed intraoperatively.

Have their anonymized ROTEM data reviewed independently by:

A panel of 3 clinical experts. AI models (ChatGPT and Gemini) using standardized prompts and ROTEM interpretation guidelines.

DETAILED DESCRIPTION:
Rotational thromboelastometry (ROTEM) is a point-of-care viscoelastic testing method used to assess the coagulation status of patients undergoing high-risk surgical procedures, such as cardiac surgery and liver transplantation. While ROTEM-guided transfusion algorithms have improved clinical outcomes, the accurate interpretation of ROTEM results remains complex and heavily dependent on clinical experience.

This prospective observational validation study aims to assess the accuracy and clinical decision-making performance of artificial intelligence (AI)-based language models in interpreting ROTEM findings. The study will compare the AI-based evaluations to expert consensus in terms of both diagnostic accuracy and treatment recommendations.

De-identified ROTEM case data will be converted into structured clinical vignettes, which will be independently interpreted by at least three experienced clinicians (serving as the gold standard) and AI models. Each AI system will be prompted with ROTEM parameters in a standardized format and asked to assess coagulopathy type and suggest appropriate treatment options. ROTEM interpretation algorithms, such as Görlinger's protocol, will be provided as background context to ensure consistent guidance.

The study will include adult patients (≥18 years) undergoing elective cardiac surgery or liver transplantation, provided complete and technically valid ROTEM results are available. The main outcome of the study is the agreement between AI-based and expert decisions regarding the need for treatment. Secondary outcomes include diagnostic classification of coagulopathy, concordance in treatment recommendations, and standard accuracy metrics (sensitivity, specificity, PPV, NPV, overall accuracy, and Cohen's Kappa).

This study does not involve any direct patient interventions or changes in treatment based on AI output. All data will be anonymized before analysis, and informed consent will be obtained from all participants.

As part of the AI evaluation and expert comparison, each ROTEM clinical scenario will be assessed based on a standardized set of 14 structured clinical questions. These questions are designed to determine both the presence and type of coagulopathy, as well as the appropriate treatment recommendations. The specific questions are:

Is there evidence of coagulopathy based on the ROTEM findings?

Do the ROTEM results indicate hyperfibrinolysis?

Do the findings suggest the presence of residual heparin effect?

Is there evidence of fibrinogen deficiency?

Is there evidence of thrombocytopenia or platelet dysfunction?

Do the results indicate coagulation factor deficiency?

Do the findings suggest protamine overdose?

Is treatment not required at this time?

Is antifibrinolytic therapy indicated?

Should protamine be administered?

Should fibrinogen or fibrinogen-containing products be administered?

Should platelet transfusion be performed?

Should prothrombin complex concentrate (PCC) or fresh frozen plasma (FFP) be administered?

If bleeding continues, should reassessment be done after 10-15 minutes?

Each question will be answered as "Yes" or "No" by both the AI system and the expert panel, and the responses will be used to calculate diagnostic and treatment concordance metrics.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing elective cardiac surgery (CABG, valve surgery, aortic procedures)
* Adult patients undergoing liver transplantation
* Availability of complete ROTEM results (EXTEM, INTEM, FIBTEM, +/- HEPTEM, APTEM)
* Informed written consent obtained

Exclusion Criteria:

* Incomplete or technically invalid ROTEM data
* Pediatric patients (<18 years)
* Refusal to participate or lack of informed consent
* Emergency and redo surgeries

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (aged 18 years and older) undergoing elective cardiac surgeries-including coronary artery bypass grafting (CABG), valve surgery, and aortic procedures-and elective liver transplantation procedures. All participants will have complete and analyzable intraoperative ROTEM (Rotational Thromboelastometry) data available. Only patients who are able to provide written informed consent will be enrolled. Emergency cases, pediatric patients, and those with technically invalid ROTEM results will be excluded.
Sampling Method: Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-05 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
treatment | 1 hour
  Agreement (yes/no) between AI model and expert panel on whether treatment is indicated.

SECONDARY OUTCOMES:
Agreement on Type of Coagulopathy as Determined by ROTEM Analysis Between AI Model and Expert Panel | 1 Hour
  Agreement on type of coagulopathy
Concordance of ROTEM-Based Treatment Recommendations Between AI and Expert Panel | 1 Hour
  Concordance of treatment recommendations (fibrinogen, PCC, plasma, protamine, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Burhan Dost, Assoc. Prof., Principal Investigator — Ondokuz Mayıs University
Locations (2):
- Turkey (Türkiye) (2):
  - İstanbul Aydın Üniversitesi Sağlık Uygulama ve Araştırma Merkezi Medical Park Florya Hastanesi, Istanbul
  - Ondokuz Mayis University, Samsun

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including demographic characteristics, surgical category, and ROTEM parameter values, may be shared upon reasonable request and at the discretion of the corresponding author. Requests will be evaluated based on the scientific validity of the proposal and availability of resources. No personal identifiers will be included, and data will be provided only after the publication of study results.
Supporting Information: Study Protocol, SAP
Time Frame: 2 years